CLINICAL TRIAL: NCT00969787
Title: DWP05195 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Daewoong Pharmaceutical Co. LTD., Daewoong Pharmaceutical Co. LTD
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: DWP05195-P001
Record Dates: First submitted 2009-07-13; First posted 2009-09-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2009-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DWP05195 (Experimental)
  Interventions: Drug: DWP05195

INTERVENTIONS:
Drug: DWP05195 — tablets, oral administration, single and multiple administrations

SUMMARY:
The purpose of this study is to evaluate safety, tolerability, pharmacokinetics and pharmacodynamics of orally administrated DWP05195 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects aged 20 to 45 years
* The subject has a Body weight ≥ 50 kg and < 90 kg and Body Mass Index (BMI) ≥ 19.0 kg/m2 and < 27.0 kg/m2
* A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints
* A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)

Exclusion Criteria:

* A subject with sign or symptoms or previously diagnosed disease of respiratory, cardiovascular, endocrinology, liver, kidney, gastrointestinal, hematology, neurology and psychology function or other significant diseases and history or suspicion of current drug abuse and alcohol abuse
* A subject who had any allergic history to any drug (prescription drug or OTC medication etc.)
* A subject who had received treatment with below listed drug within specified period prior to the first dose of study medication

  * Within last 1 month: drug or food known CYP1A2 inducer or inhibitor
  * Within 2 weeks: Prescribed or herbal or Non-prescribed medicine
  * Within 3 days: Consumption of grapefruit juice/grapefruit containing products or orange juice/orange containing products, garlic extracted functional foods
  * Within 3 days: Consumption of alcohol or caffeine
* A subject who had participated in any other clinical study within the last 12 weeks
* A subject from whom over 400mL of blood was sampled(whole blood or plasma donation, etc.) within last 12 weeks
* A Subject with the known evidence of the following infections or drug abuse
* HIV, HBs, HCV
* cannabinoid, opioid, amphetamine, cocaine, barbiturate, benzodiazepine
* Smoker or smoking cessation within 1 month or ex-smoker with positive results by cotinine test
* AST or ALT greater than 1.5 times the upper limit of reference range or QTc > 430 msec base on screening results
* Blood pressure: SBP ≥ 140 mmHg, DBP ≤ 85 mmHg
* A subject judged ineligible by the investigator to participate in this study for other reason containing clinical laboratory tests

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety & tolerability: Adverse events, vital signs, 12-Lead ECG, laboratory safety variables and physical examination | 72hr after drug administration

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax, tmax, AUC, and t½ in plasma / amount of drug, fraction, and CLr in urine Pharmacodynamics: Thermal NeuroSensory Analyser | 72 hr after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea